CLINICAL TRIAL: NCT06943235
Title: A Prospective, Multicenter, Randomized Controlled, Phase II Study of Probiotics Combined With Concurrent Hyperfractionated ChemoRadiotherapy and Adebrelimab Immunomaintenance in the Treatment of Limited-stage Small Cell Lung Cancer (LS-SCLC)
Brief Title: Study of Probiotics Combined With Concurrent Hyperfractionated ChemoRadiotherapy and Adebrelimab Immunomaintenance in the Treatment of Limited-stage Small Cell Lung Cancer (LS-SCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xingwen Fan, associate professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2503317-7
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — Probiotics; Immunotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics Combined with Concurrent Hyperfractionated Radiotherapy and Adebrelimab Immunomaintenance (Experimental): Chest radiotherapy (PTV-G: 54Gy/30F, bid; PTV-C: 45Gy/30F, bid) started before the fourth etoposide and cisplatin chemotherapy, and the subjects will be given probiotics before radiotherapy. Adebrelimab (1200mg) was given in the first week after radiotherapy, and mantained every 3 weeks for 2 year.
  Interventions: Drug: Probiotics; Radiation: concurrent Hyperfractionated Radiotherapy; Drug: Immunotherapy
- Concurrent Hyperfractionated Radiotherapy and Adebrelimab Immunomaintenance (Placebo Comparator): Chest radiotherapy (PTV-G: 54Gy/30F, bid; PTV-C: 45Gy/30F, bid) started before the fourth etoposide and cisplatin chemotherapy. Adebrelimab (1200mg) was given in the first week after radiotherapy, and mantained every 3 weeks for 2 year.
  Interventions: Radiation: concurrent Hyperfractionated Radiotherapy; Drug: Immunotherapy

INTERVENTIONS:
Drug: Probiotics — Subjects received probiotics before radiotherapy
  Arms: Probiotics Combined with Concurrent Hyperfractionated Radiotherapy and Adebrelimab Immunomaintenance
Radiation: concurrent Hyperfractionated Radiotherapy — Increase radiation dose on the basis of conventional radiotherapy
Drug: Immunotherapy — Adebrelimab, 1200mg，q3w，2 year

SUMMARY:
ADRIATIC study explored the benefits of immune maintenance therapy after LS-SCLC radiotherapy and chemotherapy. In the presence of immunotherapy, is it necessary to increase the dosage of radiotherapy and can it further improve the efficacy? This study aims to explore the efficacy and safety of simultaneous integrated boost hyperfractionation radiotherapy combined with probiotics and Adalberg monoclonal antibody consolidation therapy for small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before implementing any experimental procedures;
2. Age range: 18-80 years old;
3. Pathological diagnosis of small cell lung cancer;
4. Limited stage;
5. ECOG PS 0-1；
6. Receive ≤ 2 rounds of chemotherapy or chemotherapy plus immunotherapy;
7. Expected survival time>3 months;

Exclusion Criteria:

1. Progress after 2 induction treatments;
2. Severe emphysema, interstitial changes in the lungs, COPD patients;
3. Resting blood oxygen<93;
4. Have a history of other malignant tumors and have received chemotherapy in the past 3 years;
5. History of chest radiotherapy;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
one year progression free survival rate | one year
Complete response rate at the end of radiotherapy for one month | at the end of radiotherapy for one month

SECONDARY OUTCOMES:
One year overall survival rate | one year
one year Survival rate without distant metastasis | one year
Adverse reactions | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China